CLINICAL TRIAL: NCT03479762
Title: In Market Utilisation of Liraglutide Used for Weight Management in the UK: a Study in the CPRD Primary Care Database
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN8022-4246; U1111-1185-3276 (Other: WHO); EUPAS23369 (Registry Identifier: EU PAS Register)
Record Dates: First submitted 2018-03-21; First posted 2018-03-27 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — Liraglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Liraglutide: Patients in the CPRD primary care database who have been prescribed liraglutide after the UK launch of Saxenda® (and have no liraglutide prescriptions in the previous 12 months)
  Interventions: Drug: Liraglutide

INTERVENTIONS:
Drug: Liraglutide — No treatment given

SUMMARY:
This study is conducted in Europe. The aim of this study is to investigate the usage of liraglutide for weight management in clinical practice using the CPRD (Clinical Practice Research Datalink) primary care database.

ELIGIBILITY:
Inclusion Criteria:

-New initiators of liraglutide (unbranded, or branded prescription, i.e. Saxenda® or Victoza®), who have no liraglutide prescriptions in the twelve months prior to index date (time of first prescription). Patients must be research standard (registered as "acceptable" in the database) with at least one year of up-to-standard registration prior to their index date

Exclusion Criteria:

-Not applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in the CPRD primary care database who have been prescribed liraglutide after the UK launch of Saxenda® (and have no liraglutide prescriptions in the previous 12 months)
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2022-09-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with a BMI above or equal to 30 kg/m^2 (Saxenda® only) | Less than 6 months before the date of the first prescription
  Number
Number of patients with a BMI above or equal to 27 kg/m^2 and below 30 kg/m^2 and 1 or more comorbidities (Saxenda® only) | Less than 6 months before the date of the first prescription
  With at least 1 relevant comorbidity: (Dysglycaemia, hypertension, dyslipidaemia, obstructive sleep apnoea and/or other weight related comorbidities)
Number of patients with a BMI above or equal to 27 kg/m^2 and less than 30 kg/m^2 and no comorbidities (Saxenda® only) | Less than 6 months before the first prescription
  None of the relevant comorbidities: (Dysglycaemia, hypertension, dyslipidaemia, obstructive sleep apnoea and/or other weight related comorbidities)
Number of patients with BMI below 27 kg/m^2 (Saxenda® only) | Less than 6 months before the first prescription
  Number
Number of patients with less than 5% weight loss and continuing treatment (Saxenda® only) | Week 0 (first prescription) to week 16; week 24
  Number
Mean weight loss in patients not treated according to stopping rule (Saxenda® only) | Week 0 (first prescription) to week 16; week 24
Number of patients with a BMI not measured (Saxenda® only) | Less than 6 months before the first prescription
  Number
Number of patients with at least 5% weight loss and continuing treatment (Saxenda® only) | Week 16 - week 24
  Number

SECONDARY OUTCOMES:
Number of patients fulfilling at least one of the following: 1) a prescription interval corresponding to a daily dose of 3.0 mg, 2) dose information of 3.0 mg per day, or 3) indication of weight management (Victoza® only) | Within 4-12 weeks from the date of the first prescription
  Number of patients with Victoza® prescriptions
Number of initiators with other GLP-1 receptor agonists prescribed during continued treatment with Saxenda® (Saxenda® only) | From date of first prescription until 24 months
  Continued treatment is defined as no gaps of more than 30 days between assumed prescription end and the subsequent prescription date
Number of initiators with other products for weight management prescribed during continued treatment with Saxenda® (Saxenda® only) | From date of first prescription until 24 months
  Continued treatment is defined as no gaps of more than 30 days between assumed prescription end and the subsequent prescription date
Number of patients who have reached 3.0 mg (Saxenda® only) | 12 weeks from time of first prescription
  Number
Number of patients with a treatment duration of 0-6 months (Saxenda® only) | Month 6
  Number
Number of patients with a treatment duration of 7-12 months (Saxenda® only) | Month 12
  Number
Number of patients with a treatment duration of 13-18 months (Saxenda® only) | Month 18
  Number
Number of patients with a treatment duration of 19-24 months (Saxenda® only) | Month 24
  Number
Number of patients with a treatment duration of 25-36 months (Saxenda® only) | Month 36
  Number
Number of patients with a treatment duration of 37-48 months (Saxenda® only) | Month 48
  Number
Number of patients with a treatment duration of 49-60 months (Saxenda® only) | Month 60
  Number
Number of patients with ongoing treatment (current users) (Saxenda® only) | Month 60
  Number

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Office (2834), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Soeborg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com